CLINICAL TRIAL: NCT05811520
Title: Comparison of Scapular Stabilization and Thoracic Extension Exercises in Patients With Scapular Dyskinesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/MS-PT/01486 Maryam Qaiser
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Scapular Dyskinesis
Keywords: scapular stabilization; thoracic extension; scapular rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular stabilization exercises with conventional therapy (Experimental): The patient will sit on the knees in 90° flexion position, and a Swiss ball will be placed between the chest and stomach. From the side, the earlobe, acromion of scapula, and pelvis should made a straight line. Four general exercises will be included with 2 sets of 15 repetitions, holding for 10 sec.
  Interventions: Other: Scapular stabilization exercises with conventional therapy
- Thoracic extension exercises with conventional therapy (Experimental): Thoracic extension exercises consist of three exercise types
  Interventions: Other: Thoracic extension exercises with conventional therapy

INTERVENTIONS:
Other: Scapular stabilization exercises with conventional therapy — The patient will sit on the knees in 90° flexion position, and a Swiss ball will be placed between the chest and stomach. From the side, the earlobe, acromion of scapula, and pelvis should made a straight line. Four general exercises will be included with 2 sets of 15 repetitions, holding for 10 sec
  Arms: Scapular stabilization exercises with conventional therapy
Other: Thoracic extension exercises with conventional therapy — Thoracic extension exercises consist of three exercise protocols
  Arms: Thoracic extension exercises with conventional therapy

SUMMARY:
Scapular dyskinesis is defined as a visible alteration in scapular movement and position during rest or while performing dynamic motions causing a breakage in kinetic chain. Kinematic studies in subjects with scapular dysfunction showed decrease posterior tilt of scapula, increased scapular upward rotation and changes in glenohumeral to scapulothoracic ratios. Scapular dyskinesis can be categorized into 3 types according to standard classification. Type I is the posterior displacement of infero-medial angle due to excessive anterior tilt in sagittal plane, type II is the displacement of entire medial angle from posterior thorax caused by excessive internal rotation and dysrhythmic movement of scapula excessive elevation of superior border during scapular elevation is distinguished as type III . Almost 90% of office workers presenting with scapular and neck complains present with scapular dyskinesis . Shoulder dysfunction occur in up to 68% of individuals presenting with scapular dyskinesis

DETAILED DESCRIPTION:
Specific treatment of scapular dyskinesis include moist heat packs, soft tissue mobilization, strength and flexibility exercises of scapular muscles along with postural re-education. Acknowledging the role of scapula in upper extremity functions, integration of scapular stabilization exercises is shown to be more efficient than strengthening and stretching exercises for enhancing shoulder proprioception, optimizing muscle strength and decreasing dyskinesis. Scapular stabilization exercises defined as exercises aimed at gaining stability and strength of scapular muscles and increasing neuromuscular control to maintain the proper position of the scapula.

These exercises increase fiber strength, mass, capillaries volume thus increasing the blood flow of muscle.

Mobility of Thoracic spine is an important factor to consider while treating scapular dyskinesis as reduced thoracic mobility can result in dramatic reduction of shoulder range of motion

. So a rehabilitation protocol based on the scapula dynamic stability to restore the position, direction and movement pattern of scapula by stabilizing and retraining the scapular muscles is a possible intervention strategy for improving recovery and preventing shoulder dysfunction. Numerous exercises had been proposed for rehabilitation of dyskinesis, but it lack consensus on which exercise is effective in each type of dyskinesia. As different types of scapular dyskinesia have different manifestations of muscle imbalance

ELIGIBILITY:
Inclusion Criteria:

* > 1.5 cm difference on lateral scapular slide test
* Ability to perform shoulder abduction at neutral position
* Presence of any type of scapular dyskinesis
* Asymmetrical scapular position at rest or winging seen during inspection of scapula
* Patients volunteered to participate in the study and signed informed consent

Exclusion Criteria:

* Patients with Structural scoliosis
* Patients with secondary conditions (Neoplasm, Neurological or vascular disorders)
* Patient undergone surgical treatment of shoulder or upper limb
* Patient with disc prolapse, spinal stenosis and fibromyalgia
* Infectious or inflammatory arthritis of spine
* Severe bone conditions (osteoporosis)
* Psychosocial disturbances

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
inclinometer | four weeks
  Used to measure the scapular posterior tilt (type I dyskinesis), external rotation (type II dyskinesis) and upward rotation (type III dyskinesis) at different humeral abduction and flexion angles. The starting position was the elbow extension and wrist neutral position in the standing pose. Inclinometer is brought into contact with the scapula spine and scapular movements were measured at different angles.
vernier calliper | four weeks
  Used to evaluate the scapular index (indicator of position of scapula in static pose). The Scapular Index value is calculated using the following equation:
  Scapular Index = [(distance from the sternal notch to the coracoid process/distance from the posterolateral angle of the acromion to the third spinous process of the thoracic spine) × 100]
goniometer | four weeks
  Universal goniometer for range of motion measurement of shoulder joint.
Disability of the Arm, Shoulder, and Hand Outcome Questionnaire | four weeks
  The Disability of the Arm, Shoulder, and Hand Outcome Questionnaire evaluation tool consists of total of 30 items, scored on a five-point scale (no difficulty, slightly difficult, moderately difficult, very difficult, or not at all).

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No